CLINICAL TRIAL: NCT00636246
Title: Sertraline/[S,S]-Reboxetine Combination Versus Sertraline And [S,S]-Reboxetine Monotherapy In Major Depressive Disorder (MDD) In A Double-Blind, Placebo-Controlled, Eight Week Study.
Brief Title: A Comparison of Sertraline-reboxetine Combination Therapy Versus Sertraline or Reboxetine Monotherapy in the Treatment of Major Depression.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0501075
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Sertraline/[S,S]-Reboxetine-satellite150/4 (Experimental)
  Interventions: Drug: sertraline/[S,S]-reboxetine
- Sertraline/[S,S]-Reboxetine-satellite150/6 (Experimental)
  Interventions: Drug: sertraline/[S,S]-reboxetine
- sertraline-satellite (Active Comparator)
  Interventions: Drug: sertraline
- sertraline-main (Active Comparator)
  Interventions: Drug: sertraline
- Sertraline/[S,S]-Reboxetine-satellite150/2 (Experimental)
  Interventions: Drug: sertraline/[S,S]-reboxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Sertraline/[S,S]-Reboxetine-main (Experimental)
  Interventions: Drug: sertraline/[S,S]-reboxetine
- [S,S]-reboxetine-main (Active Comparator)
  Interventions: Drug: [S,S]-reboxetine monotherapy

INTERVENTIONS:
Drug: sertraline/[S,S]-reboxetine — Tablets, 50mg sertraline/2mg [S,S]-reboxetine for 3 days orally, followed by 100mg sertraline/4mg [S,S]-reboxetine for 4 and one half weeks, followed by 150mg sertraline/4mg [S,S]-reboxetine for 5 and one half weeks.
  Arms: Sertraline/[S,S]-Reboxetine-satellite150/4
Drug: sertraline/[S,S]-reboxetine — Tablets, 50mg sertraline/2mg [S,S]-reboxetine for 3 days orally, followed by 100mg sertraline/4mg [S,S]-reboxetine for 4 and one half weeks, followed by 150mg sertraline/6mg [S,S]-reboxetine for 5 and one half weeks.
  Arms: Sertraline/[S,S]-Reboxetine-satellite150/6
Drug: sertraline — Tablets, 50 mg/day orally for 3 days, followed by 100 mg/day orally for 4 and one half weeks, followed by 150 mg/day orally for 3 weeks.
  Arms: sertraline-satellite
Drug: sertraline — Tablets, 50 mg/day orally for 3 days, followed by 100 mg/day orally for 4 and one half weeks, followed by 150 mg/day orally for 3 weeks
  Arms: sertraline-main
Drug: sertraline/[S,S]-reboxetine — Tablets, 50mg sertraline/2mg [S,S]-reboxetine for 3 days orally, followed by 100mg sertraline/2mg [S,S]-reboxetine for 4 and one half weeks, followed by 150mg sertraline/2mg [S,S]-reboxetine for 5 and one half weeks.
  Arms: Sertraline/[S,S]-Reboxetine-satellite150/2
Drug: Placebo — Tablets, orally once per day for 8 weeks
  Arms: Placebo
Drug: sertraline/[S,S]-reboxetine — Tablets, 50mg sertraline/2mg [S,S]-reboxetine orally for 3 days, followed by 100mg sertraline/2mg [S,S]-reboxetine for 4 and one half weeks, followed by 150mg sertraline/2mg [S,S]-reboxetine for 5 and one half weeks
  Arms: Sertraline/[S,S]-Reboxetine-main
Drug: [S,S]-reboxetine monotherapy — Tablets, 2 mg/day orally for 3 days, followed by 4 mg/day orally for 4 and one half weeks, followed by 6mg/day for 3 weeks
  Arms: [S,S]-reboxetine-main

SUMMARY:
This study was designed to determine if the novel combination of the SSRI, sertraline, and the NRI reboxetine will increase antidepressant efficacy without sacrificing the favorable safety profile of SSRIs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must fulfill the criteria for MDD without psychotic features as defined by DSMIV, based on clinical assessment and confirmed by Structural Clinical Interview for DSM-IV Axis I Disorder-Clinical Version (SCID-I) plus the MDD Specifiers included in the Research Version of SCID-I.
* HAM-D (17-item) ≥ 22 at Screening (Visit 1) and > 20 at Baseline (Visit 2).
* Minimum CGI-S ≥ 4 at Screening (Visit 1) and at Baseline (Visit 2).

Exclusion Criteria:

* Known failure to satisfactory respond after adequate dose and duration (12 weeks) of treatment with clomipramine and one SSRI, or with two or more SSRIs.
* Subjects with > 20% HAM-D (17-item) improvement (decrease) from Screening (Visit 1) at Baseline (Visit 2).
* Subjects with uncorrected hypothyroidism or hyperthyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2004-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The change from Baseline up to Week 8 (Visit 9) in the Montgomery-Asberg Depression Rating Scale (MADRS) total score as measured by a mixed concentration, suicidal ideation and restlessness. | visits 1-9

SECONDARY OUTCOMES:
Change from Baseline in HAM-D (17-item) total score | Weeks 1, 2, 3, 5, 6, and 8
Change from Baseline in the Hamilton Anxiety Rating Scale (HAM-A) and Apathy Evaluation Scale (AES) | Weeks 5 and 8
The frequency and severity of treatment-emergent adverse events, ECG changes, laboratory and vital signs changes by treatment group using descriptive statistics. | Weeks 1, 2, 3, 5, 6, and 8
Change from Baseline in MADRS total score | Weeks 1, 2, 3, 5, 6, and 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Estonia (4):
  - Pfizer Investigational Site, Viljandi, Viljandi Mk.
  - Pfizer Investigational Site, Pärnu
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Russia (6):
  - Pfizer Investigational Site, Kazan'
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Rostov-on-Don
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk
  - Pfizer Investigational Site, Tomsk

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501075&StudyName=A%20comparison%20of%20sertaline-reboxetine%20combination%20therapy%20versus%20sertaline%20or%20reboxatine%20monotherapy%20in%20the%20treatment%20of%20major%20depression.